CLINICAL TRIAL: NCT00839852
Title: A Long-term, Open-label Extension Study of the Safety and Tolerability of RGH-188 (Cariprazine) in Patients With Schizophrenia
Brief Title: A Study of Cariprazine in Patients With Chronic Stable Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGH-MD-17
Record Dates: First submitted 2009-02-05; First posted 2009-02-10 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — cariprazine

ARMS (1):
- Cariprazine 1.5mg (Experimental): Participants received cariprazine 1.5 mg capsule once, twice or three times a day depending on their response and tolerability
  Interventions: Drug: Cariprazine

INTERVENTIONS:
Drug: Cariprazine — Cariprazine was supplied in capsules.
  Other Names: RGH-188

SUMMARY:
This is an outpatient study to evaluate the long-term safety, tolerability, and pharmacokinetics of cariprazine in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed the double-blind treatment period of the lead-in study RGH-MD-16 (NCT 00694707)
* Patients who have responded to double-blind treatment in the lead-in study as defined as ≥ 20% reduction relative to Visit 2 (Baseline) of the Positive and Negative Syndrome Scale (PANSS) total score and a Clinical Global Impressions-Severity (CGI-S) score of ≤ 3.
* Patients eligible to continue as outpatients based on the opinion of the Principal Investigator.
* Patients must have a caregiver to ensure treatment compliance.

Exclusion Criteria:

* Patients with clinically significant abnormalities on physical examination, laboratory, vital signs, and/or electrocardiogram (ECG).

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2009-05-31 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2010-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Durgam, MD, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories, Inc.
Locations (57):
- United States (17):
  - Forest Investigative Site, Costa Mesa, California
  - Forest Investigative Site, Long Beach, California
  - Forest Investigative Site, Oceanside, California
  - Forest Investigative Site, Paramount, California
  - Forest Investigative Site, Riverside, California
  - Forest Investigative Site, Washington D.C., District of Columbia
  - Forest Investigative Site, Bradenton, Florida
  - Forest Investigative Site, Kissimmee, Florida
  - Forest Investigative Site, Lake Charles, Louisiana
  - Forest Investigative Site, Baltimore, Maryland
  - Forest Investigative Site, Flowood, Mississippi
  - Forest Investigative Site, Creve Coeur, Missouri
  - Forest Investigative Site, Cincinnati, Ohio
  - Forest Investigative Site, Charleston, South Carolina
  - Forest Investigative Site, Memphis, Tennessee
  - Forest Investigative Site, Houston, Texas
  - Forest Investigative Site, Irving, Texas
- India (12):
  - Forest Investigative Site, Vijaywada, Andh Prad
  - Forest Investigative Site, Visakhapatnam, Andh Prad
  - Forest Investigative Site, Ahmedabad, Gujarat
  - Forest Investigative Site, Bangalore, Karna
  - Forest Investigative Site, Mangalore, Karna
  - Forest Investigative Site, Manipal, Karna
  - Forest Investigative Site, Mysore, Karna
  - Forest Investigative Site, Pune, Mahara
  - Forest Investigative Site, Jaipur, Rajasthan
  - Forest Investigative Site, Chennai, Tamil Nadu
  - Forest Investigative Site, Tirupati, Tamil Nadu
  - Forest Investigative Site, Kanpur, Uttar Prad
- Malaysia (3):
  - Forest Investigative Site, Johor Bahru
  - Forest Investigative Site, Kuala Lumpur
  - Forest Investigative Site, Perak
- Russia (15):
  - Forest Investigative Site, Arkhangelsk
  - Forest Investigative Site, Gatchina
  - Forest Investigative Site, Ivanovo
  - Forest Investigative Site, Kazan'
  - Forest Investigative Site, Krasnodar
  - Forest Investigative Site 204, Moscow
  - Forest Investigative Site 206, Moscow
  - Forest Investigative Site, Moscow
  - Forest Investigative Site, Nizhny Novgorod
  - Forest Investigative Site 214, Saint Petersburg
  - Forest Investigative Site 217, Saint Petersburg
  - Forest Investigative Site, Saint Petersburg
  - Forest Investigative Site 202, Saint Petersburg
  - Forest Investigative Site 203, Saint Petersburg
  - Forest Investigative Site, Samara
- Ukraine (10):
  - Forest Investigative Site, Kherson, Vil. Stepanivka
  - Forest Investigative Site, Chernihiv
  - Forest Investigative Site, Dnipropetrovsk
  - Forest Investigative Site, Donetsk
  - Forest Investigative Site, Hlevakha
  - Forest Investivative Site, Kharkiv
  - Forest Investigative Site, Kiev
  - Forest Investigative Site, Kyiv
  - Forest Investigative Site, Odesa
  - Forest Investigative Site, Ternopil

REFERENCES:
- [Derived] Laszlovszky I, Barabassy A, Nemeth G. Cariprazine, A Broad-Spectrum Antipsychotic for the Treatment of Schizophrenia: Pharmacology, Efficacy, and Safety. Adv Ther. 2021 Jul;38(7):3652-3673. doi: 10.1007/s12325-021-01797-5. Epub 2021 Jun 6. PMID 34091867
- [Derived] Barabassy A, Sebe B, Acsai K, Laszlovszky I, Szatmari B, Earley WR, Nemeth G. Safety and Tolerability of Cariprazine in Patients with Schizophrenia: A Pooled Analysis of Eight Phase II/III Studies. Neuropsychiatr Dis Treat. 2021 Apr 7;17:957-970. doi: 10.2147/NDT.S301225. eCollection 2021. PMID 33854317
- [Derived] Nasrallah HA, Earley W, Cutler AJ, Wang Y, Lu K, Laszlovszky I, Nemeth G, Durgam S. The safety and tolerability of cariprazine in long-term treatment of schizophrenia: a post hoc pooled analysis. BMC Psychiatry. 2017 Aug 24;17(1):305. doi: 10.1186/s12888-017-1459-z. PMID 28836957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Enrolled Population consisted of 97 participants who completed the lead-in study, RGH-MD-16, and signed an informed consent form to continue in this extension study.
  The Safety Population consisted of 93 participants from the Enrolled Population who took at least 1 dose of cariprazine in this extension study.
Pre-assignment Details: The study was designed as a one-arm study where patients were not randomized or analyzed by dose, rather they were flexibly dosed with Cariprazine 1.5, 3.0, or 4.5 mg/day via oral administration. The starting dose of 1.5 mg/day was titrated as needed within the range of 1.5-4.5 mg/d based on investigator's judgment of response and tolerability.
Groups:
- Cariprazine: Participants received cariprazine 1.5 mg capsule once, twice or three times a day depending on their response and tolerability
Period: Overall Study
Arm/Group | Cariprazine
Started | 93
Completed | 46
Not Completed | 47
Not completed — Adverse Event | 10
Not completed — Insufficient Therapeutic Response | 3
Not completed — Protocol Violation | 9
Not completed — Withdrawal of Consent | 16
Not completed — Lost to Follow-up | 7
Not completed — Lack of Compliance While in Jail | 1
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Population: Safety population: All enrolled participants who took at least 1 dose of cariprazine.
Arm/Group | Cariprazine
Number analyzed (Participants) | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 88
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 30
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 52
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 72.19 (17.66)
Height [Mean (Standard Deviation); unit: cm] | 169.09 (10.73)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.99 (4.46)
Waist circumference [Mean (Standard Deviation); unit: cm] | 84.90 (11.19)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 48 in the PANSS Total Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a 30-item rating scale that assesses the positive and negative symptoms of individuals with schizophrenia. Responses to the 30 items are based on a structured clinical interview with the patient and on supporting clinical information obtained from family, hospital staff, or other reliable informants. Of the 30 psychiatric parameters measured by the scale, 7 assess positive symptoms (eg, delusions, grandiosity); 7 assess negative symptoms (eg, blunted affect, emotional withdrawal); and 16 assess general psychopathology (eg, poor attention, active social avoidance). Each item is scored on a 7-point scale (1 = absent, 2 = minimal, 3 = mild, 4 = moderate, 5 = moderately severe, 6 = severe, and 7 = extreme). The PANSS total score can range from 30 to 210. A higher score indicates worse symptoms. A negative change score indicates improvement.
Time Frame: Baseline to Week 48
Population: Intent-to-treat population: All participants who took at least 1 dose of cariprazine and who had at least 1 post-baseline assessment of the PANSS total score.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Cariprazine
Number analyzed (Participants) | 92
Units on a scale | -38.5 (1.5)

2. Secondary Outcome: Change From Baseline to Week 48 in the CGI-S Score
Description: The Clinical Global Impressions-Severity (CGI-S) scale is a 7-point scale that measures the overall severity of the illness compared with the severity of illness in other patients the Investigator has observed. The Investigator assesses the severity of the patient's illness as one of the following: 1 = Normal, not at all ill; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill patients. The CGI-S score can range from 1 to 7. A higher score indicates more severe illness. A negative change score indicates improvement.
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Cariprazine
Number analyzed (Participants) | 92
Units on a scale | -2.0 (0.1)

ADVERSE EVENTS:
Time Frame: Baseline to Week 52
Description: Safety population: All enrolled participants who took at least 1 dose of cariprazine.
Arm/Group | Cariprazine
All-Cause Mortality (participants affected / at risk) | 0/93
Serious Adverse Events (participants affected / at risk) | 12/93
Other Adverse Events (participants affected / at risk) | 62/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cariprazine (N=93)
Schizophrenia (Psychiatric disorders) | 4
Psychotic disorder (Psychiatric disorders) | 2
Adjustment disorder (Renal and urinary disorders) | 1
Agitation (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Social stay hospitalisation (Social circumstances) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Filariasis (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cariprazine (N=93)
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 5
Nasopharyngitis (Infections and infestations) | 8
Weight increased (Investigations) | 11
Akathisia (Nervous system disorders) | 13
Headache (Nervous system disorders) | 8
Dizziness (Nervous system disorders) | 7
Tremor (Nervous system disorders) | 7
Extrapyramidal disorder (Nervous system disorders) | 6
Sedation (Nervous system disorders) | 5
Somnolence (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 13
Agitation (Psychiatric disorders) | 7
Anxiety (Psychiatric disorders) | 7
Psychotic disorder (Psychiatric disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.